CLINICAL TRIAL: NCT03384160
Title: Evaluation of Articaine 4% Versus Mepivacaine 2% for Surgery of Molars Thirds: Splint-mouth Randomized Double Blind Controlled Clinical Trial.
Brief Title: Evaluation of Articaine 4% Versus Mepivacaine 2% for Surgery of Molars Thirds: Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Prof. Dr. Fernando Vagner Raldi (Unknown); Paula Carolina de Almeida (Unknown)
Responsible Party: Principal Investigator, Michelle Bianchi de Moraes, Assistant Professor, Department of Diagnosis and Surgery, São Paulo State University (Unesp), Institute of Science and Technology, São José dos Campos, Brazil., Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ICT-UNESP
Record Dates: First submitted 2017-12-17; First posted 2017-12-27 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Pain; Teeth, Impacted
Keywords: Pain; Third molar; Articaine; Mepivacaine
MeSH Terms: conditions — Pain; Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: The sample will consist of 32 lower third molars, semi-inclusively or included. This study will be a randomized, double blind, controlled, split-mouth clinical trial, divided into two groups simultaneously, namely:
  Group 1 (16 teeth) - using anesthetic mepivacaine in third molar extraction. Group 2 (16 teeth) - using anesthetic articaine in third molar extraction
Who Masked: Participant, Care Provider
Masking Description: Surgical procedures were always performed by the same surgeon and assistant, who was unaware of the group that belonged to the patient, as well as the patient himself. This randomization was performed involving numbers and envelopes, being only the investigator's knowledge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1-Pain monitor (Active Comparator): Use of the anesthetic Mepivacaine 2% in third molar extraction
  Interventions: Diagnostic Test: Group 2 -Pain monitor
- Group 2 -Pain monitor (Active Comparator): Use of the anesthetic Articaine 4% in third molar extraction
  Interventions: Diagnostic Test: Group 1 -Pain monitor

INTERVENTIONS:
Diagnostic Test: Group 1 -Pain monitor — Use of the anesthetic Mepivacaine 2% in third molar extraction and evaluation in postoperative
  Arms: Group 2 -Pain monitor
Diagnostic Test: Group 2 -Pain monitor — Use of the anesthetic Articaine 4% in third molar extraction and evaluation in postoperative
  Arms: Group 1-Pain monitor

SUMMARY:
The extraction of third molars, a frequent treatment in clinical dental practice, can lead patients to painful symptoms during and after surgery. The dental surgeon must correctly indicate the need for extraction and also provide patients who need this treatment greater comfort and control of pain in the trans and postoperative period. Thus, it is necessary to use an effective local anesthetic favoring the factors inherent to the postoperative and achieving good treatment results.

DETAILED DESCRIPTION:
This study will compare the use of Articaine at 4% to that of Mepivacaine at 2% for lower third molar surgeries semi-included and / or included. I will select 16 patients who require surgical treatment for extraction of third molars, aged between 16 and 40 years at the São Paulo State University. These will participate simultaneously in the two groups: Group 1 mepivacaine (MEP) and Group 2 articaine (ART), and the division will be performed by randomization, so that each patient will have each side (right or left) allocated in different groups. The primary evaluation variable will be to compare the pain index in the immediate postoperative period, using Visual Analog Scale (VAS), and will also analyze Hemodynamic Parameters, such as Patient and Operator satisfaction. The results will be submitted to qualitative and quantitative statistical analysis. The descriptive data will be compared using the statistical analysis of variance (ANOVA) and Tukey test with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Classification -(ASA I) patients;
* Patients with need for extraction of lower third molars included and / or semi-included;
* Teeth in opposing hemiarch with the same classifications as Pell and Gregory and Winter;
* Age between 16 and 40 years;
* Patients who agree to voluntarily participate in the survey.

Exclusion Criteria:

* History of allergic reactions (hypersensitivity) to anesthetics;
* Patients presenting with local or systemic alterations that contraindicate the procedure;
* Current use of drugs that may interfere with the action of anesthetics;
* Need for sedatives or anxiolytic drugs during extraction;
* Pregnancy or breastfeeding;
* Third erupted lower third molars.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Pain assessment | The scale will be provided on paper and divided into postoperative hours up to 3 days.
  Evaluated in patients in groups 1 and 2. Scale of Visual Analog Scale (VAS), with values from zero to ten, being zero without pain and ten the maximum of pain. This scale will be provided on paper and divided into postoperative hours up to 3 days.

SECONDARY OUTCOMES:
Assessment of blood pressure change | Observed and recorded immediately before application of the anesthetic solution, at 5, 20 and 70 minutes after the application of anesthesia
  Evaluated in patients submitted to the exodontia of third molars, with different types of anesthetics.The investigator evaluated with auscultatory instrument.

OTHER OUTCOMES:
Assessment of heart rate change | Observed and recorded immediately before application of the anesthetic solution, at 5, 20 and 70 minutes after the application of anesthesia
  Evaluated in patients submitted to the exodontia of third molars.
Assessment of oxygen saturation change | Observed and recorded immediately before application of the anesthetic solution, at 5, 20 and 70 minutes after the application of anesthesia
  Evaluated in patients submitted to the exodontia of third molars

CONTACTS AND LOCATIONS:
Overall Officials: Michelle B Moraes, PHD, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho-Unesp
Locations (1):
- Michelle Bianchi de Moraes, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brockmann WG. Mepivacaine: a closer look at its properties and current utility. Gen Dent. 2014 Nov-Dec;62(6):70-5; quiz 76. PMID 25369391
- [Result] Colombini BL, Modena KC, Calvo AM, Sakai VT, Giglio FP, Dionisio TJ, Trindade AS Jr, Lauris JR, Santos CF. Articaine and mepivacaine efficacy in postoperative analgesia for lower third molar removal: a double-blind, randomized, crossover study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Aug;102(2):169-74. doi: 10.1016/j.tripleo.2005.09.003. Epub 2006 Mar 24. PMID 16876058
- [Result] Gregorio LV, Giglio FP, Sakai VT, Modena KC, Colombini BL, Calvo AM, Sipert CR, Dionisio TJ, Lauris JR, Faria FA, Trindade Junior AS, Santos CF. A comparison of the clinical anesthetic efficacy of 4% articaine and 0.5% bupivacaine (both with 1:200,000 epinephrine) for lower third molar removal. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Jul;106(1):19-28. doi: 10.1016/j.tripleo.2007.11.024. Epub 2008 Apr 16. PMID 18420431
- [Result] Holliday R, Jackson I. Superior position of the mandibular foramen and the necessary alterations in the local anaesthetic technique: a case report. Br Dent J. 2011 Mar 12;210(5):207-11. doi: 10.1038/sj.bdj.2011.145. PMID 21394145
- [Result] McCoy JM. Complications of retention: pathology associated with retained third molars. Atlas Oral Maxillofac Surg Clin North Am. 2012 Sep;20(2):177-95. doi: 10.1016/j.cxom.2012.06.002. No abstract available. PMID 23021395